CLINICAL TRIAL: NCT02052258
Title: Oxytocin in Opiate Dependence: A Double-blind, Within-subjects, Placebo-controlled Pilot Study of the Effects of Intranasal Oxytocin on Emotional Processes and Stress Responses in Patients With Opiate Dependence
Brief Title: Oxytocin in Opiate Dependence: A Pilot Study of the Effects of Intranasal Oxytocin on Emotional Processes and Stress Responses in Patients With Opiate Dependence
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MacDonald, Kai, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 120283
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Opiate Dependence
Keywords: oxytocin
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxytocin

ARMS (1):
- oxytocin (Experimental)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
Opiate dependence is a serious problem, and oxytocin has many properties which make it attractive as a treatment for this type of substance dependence. This experiment will test the effects of oxytocin on a variety of brain-based processes in patients with opiate dependence. The investigators hypothesize that intranasal oxytocin in these conditions will enhance emotional processing and will have beneficial effects on stress responses in opiate-dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* adult men 18 years or older
* meet DSM-IV criteria for opiate dependence, and no other active substance dependence disorder save nicotine dependence
* clinically stable, and low risk for suicide as determined by principal investigator and screening questionnaire
* abstinent from non-prescribed opiate use for at least two weeks from Baseline 1 and free from opiate withdrawal symptoms. If on agonist therapy, dose must be stable for 2 weeks before study visit.
* must be able to use nasal spray
* negative salivary drug screen, save for opiates

Exclusion Criteria:

* any active medical condition that in the opinion of the investigator will interfere with the objectives of the study
* any active, severe mental illness, neurological disorder, including schizophrenia, autism, Asperger's syndrome
* are unsuitable in any way to participate in this study, in the opinion of the investigator
* hospitalizations due to complications of an Axis 1 disorder for the past 12 months, excluding drug or alcohol rehabilitation
* any clinically significant chronic pain condition, as determined by the principal investigator
* positive salivary drug screen at the time of the visit, for any substance other than opiates or another prescribed medication

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Cold Pressor Task | up to 5 minutes
  The Cold Pressure task involves placing a hand or forearm in cold water, a stimulus that produces a slowly mounting pain of mild to moderate intensity and is terminated by voluntary withdrawal of the limb. The cold pressor task has been used in many studies of pain, autonomic reactivity, and hormonal stress responses.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Medical Center, San Diego, California, United States